CLINICAL TRIAL: NCT07093970
Title: A Phase I/II, Open-label, Multi-center, Dose Escalation and Expansion Study to Assess the Safety, Tolerability, Efficacy and Pharmacokinetics of MRG006A in Patients With Advanced Solid Tumors
Brief Title: A Study of MRG006A in the Treatment of Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lepu Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRG006A-001
Record Dates: First submitted 2025-07-22; First posted 2025-07-30 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors
Keywords: MRG006A; Antibody Drug Conjugate (ADC); Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRG006A (Experimental): All patients in Phase I and Phase II will be administrated MRG006A on Day 1 of every 3 weeks (21-day cycle).
  Interventions: Drug: MRG006A

INTERVENTIONS:
Drug: MRG006A — Administrated intravenously

SUMMARY:
The objective of this study is to assess the safety, efficacy, pharmacokinetics, and immunogenicity of MRG006A in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This study consists of two parts. Phase I is a dose escalation study to determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of MRG006A. Phase II is a dose expansion study to further assess the efficacy, safety, pharmacokinetics and immunogenicityof MRG006A at confirmed RP2D.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and provide written informed consent and comply with the requirements set forth in the protocol.
2. age ≥ 18 years, ≤ 75 years.
3. Expected survival ≥ 3 months.
4. For patients with stage I and II disease, tumor tissue samples for GPC3 and P53 testing must be provided.
5. Patients with histologically or cytologically confirmed advanced solid tumors.
6. At least one measurable lesion according to RECISTv1.1 and mRECIST (HCC patients).
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Organ function must meet basic requirements.
9. Women who are pregnant or breastfeeding are not included in this study.
10. Female and male patients of childbearing potential must agree to take adequate measures.

Exclusion Criteria:

1. Moderate and above thoracoabdominal pelvic fluid and pericardial effusion with clinical symptoms.
2. History of liver failure and hepatic encephalopathy.
3. Portal vein tumor thrombus involving both the main portal vein and left and right branches, or involving both the main portal vein and mesenteric vein needs to be excluded. The tumor involves the vena cava, or has formed a vena cava tumor thrombus.
4. Residual toxicity due to previous anti-tumor therapy or clinically significant laboratory abnormalities higher than grade 1 (CTCAEv5.0).
5. For liver cancer, previous or current central nervous system metastases and/or meningeal metastases. Patients with treated stable brain metastases from non-hepatic cancers may participate.
6. Patients at high risk of bleeding.
7. Severe cardiac insufficiency within 6 months prior to enrollment.
8. Pulmonary embolism or deep venous thrombosis within 3 months before the first study drug treatment;
9. History of gastrointestinal perforation, fistula, and bowel obstruction, extensive bowel resection, Crohn 's disease, ulcerative colitis, or chronic diarrhea for the past 6 months.
10. Patients with double cancer and multiple cancer.
11. Uncontrolled or poorly controlled disease.
12. History of ventricular tachycardia or torsades de pointes.
13. Previous or combined interstitial pneumonia, severe chronic obstructive pulmonary disease with respiratory failure, severe pulmonary insufficiency, symptomatic bronchospasm and other medical history;
14. Allergic reactions to any component or excipient of MRG006A, or known Grade ≥ 3 allergic reactions to other prior anti-GPC3 or other monoclonal antibodies.
15. Acute or chronic active hepatitis B or C infection.
16. Active or clinically poorly controlled serious infection.
17. Receiving anti-tuberculosis treatment or receiving anti-tuberculosis treatment within 1 year before the first dose.
18. People infected with human immunodeficiency virus (HIV), known syphilis infection requiring treatment.
19. Use of systemic corticosteroids within 4 weeks prior to first treatment.
20. Use of strong CYP3A4 inducers, strong CYP3A4 inhibitors within 14 days or 5 times the half-life prior to the first dose.

Ages: 17 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 343 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) - Phase I | Baseline to the end of the first treatment cycle (each cycle is 21 days).
  The highest dose confirmed wherein less than 2 out of 6, or < 33% of evaluable patients in a treatment cohort experiences dose-limiting toxicity (DLT).
Recommended Phase II Dose (RP2D) - Phase I | Baseline to study completion (up to 24 months).
  The dose level of MRG006A recommended for further clinical studies based on assessment of the safety, efficacy and PK data from this study.
Adverse Events (AEs) - Phase I | Baseline to 30 days after the last dose of study treatment.
  Any reaction, side effect, or untoward event that occurs during the course of the clinical trial whether or not the event is considered related to the study drug.
Serious Adverse Events (SAEs) - Phase I | Baseline to 30 days after the last dose of study treatment.
  Adverse events that are fatal, life-threatening, or result in hospitalization or prolonged hospitalization, persistent or significant disability/incapacity/substantial disruption of the ability to lead a normal life, congenital anomaly/birth defect or major medical events or reactions.
Objective Response Rate (ORR)- Phase II | Baseline to study completion (up to 24 months).
  ORR is defined as the proportion of subjects with CR and PR assessed by IRC and investigator according to RECIST v1.1 and mRECIST（HCC patients）. And determine the objective response rate (CR + PR) and its 95% confidence interval.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) - Phase I | Baseline to study completion (up to 24 months).
  ORR is defined as the proportion of subjects with CR and PR assessed by IRC and investigator according to RECIST v1.1 and mRECIST（HCC patients）. And determine the objective response rate (CR + PR) and its 95% confidence interval.
Overall Survive (OS)- Phase II | Baseline to study completion (up to 24 months).
  The time from start of study treatment to date of death as a result of any cause.
Duration of Response (DoR) | Baseline to study completion (up to 24 months).
  The time interval between the date of the earliest qualifying response and the date of disease progression or death for any cause, whichever occurs earlier.
Disease Control Rate (DCR) | Baseline to study completion (up to 24 months).
  The proportion of patients who achieve CR, PR, or stable disease (SD) after treatment.
Progression Free Survival (PFS) | Baseline to study completion (up to 24 months).
  The time from the date of first study dose to disease progression or death whichever occurs first.
Cmax | Baseline to 30 days after the last dose of study treatment.
  Maximum observed blood concentration
Tmax | Baseline to 30 days after the last dose of study treatment.
  Time to reach the maximum blood concentration.
AUC0-t | Baseline to 30 days after the last dose of study treatment.
  Area under the blood concentration-time curve from time 0 to the time of last quantifiable concentration.
Incidence of anti-drug antibody (ADA) | Baseline to 30 days after the last dose of study treatment.
  The proportion of patients with positive ADA results.
QT interval corrected by Fridericia's formula（QTcF） | Baseline to 15 days after the third dose of study treatment.
  Evaluate the effect of MRG006A on the prolongation of QT interval corrected by heart rate using Fridericia's formula (QTcF) in patients with advanced solid tumors.
Adverse Events (AEs) - Phase II | Baseline to 30 days after the last dose of study treatment.
  Any reaction, side effect, or untoward event that occurs during the course of the clinical trial whether or not the event is considered related to the study drug.
Serious Adverse Events (SAEs) - Phase II | Baseline to 30 days after the last dose of study treatment.
  Adverse events that are fatal, life-threatening, or result in hospitalization or prolonged hospitalization, persistent or significant disability/incapacity/substantial disruption of the ability to lead a normal life, congenital anomaly/birth defect or major medical events or reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhou, M.D., Principal Investigator — Fudan University; Hong Zhao, M.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (2):
- China (2):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No